CLINICAL TRIAL: NCT01739062
Title: Prostate Cancer Risk Assessment Using Genetic Markers in General Practice
Brief Title: The ProCaRis Study: Prostate Cancer Risk Assessment in General Practice
Acronym: ProCaRis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Velux Fonden (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2011-41-6904
Record Dates: First submitted 2012-11-27; First posted 2012-11-30 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
Keywords: PSA test; Prostate cancer; Genetic screening
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Polymorphism, Single Nucleotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Genetic risk assessment (Experimental): At least 40 SNP (single nucleotide polymorphisms)increase the risk of PCa. The individual risk of PCa accumulates with the increasing number of these genetic variants. The risk is doubled if patient has familial disposition as well. In retrospective studies, non-genetic risk-prediction models were compared to risk-prediction models containing both non-genetic factors and SNPs analyses. The genetic models had a significantly higher specificity than the non-genetic models. It has been argued that genetic PCa risk assessment could reduce the inexpedient use of PSA tests, saving it for patients at high risk of PCa.
  Interventions: Genetic: Genetic risk assessment
- Familial disposition risk assessment (No Intervention)

INTERVENTIONS:
Genetic: Genetic risk assessment
  Other Names: Single nucleotide polymorphism
  Arms: Genetic risk assessment

SUMMARY:
The preferred method for early detection of prostate cancer (PCa) in older men with family history is the Prostate Specific Antigen test (PSA test), although the method is imprecise. It produces a high number of false-positive results and increases the risk of over-diagnosis and over-treatment. Yet, an increasing number of men get the PSA test as part of unsystematic screening. Genetic risk assessment may be a better way to identify men with low risk of PCa. The main study hypothesis is that genetic information about low risk of PCa can reduce the number of patients who get a PSA test as part of unsystematic screening.

ELIGIBILITY:
Inclusion Criteria:

* patients who receive a PSA test

Exclusion Criteria:

* age over 80 years
* elevated PSA-level (> 4,0 ng/ml) concurrently or within previous 2 years
* prostate or bladder disease
* prostate cancer
* non-Caucasians
* do not speak and understand Danish

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2031-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of low risk patients who get a PSA test | 1 year, 2 years
  The primary objective of this study is to evaluate the impact on use of PSA tests of introducing genetic PCa risk assessment in general practice.

CONTACTS AND LOCATIONS:
Overall Officials: Karina D Sørensen, PhD, Principal Investigator — Department of Molecular Medicine, Aarhus University Hospital, Denmark; Flemming Bro, Professor, Study Chair — The Research Unit for General Practice, Aarhus University, Denmark; Peter Vedsted, Professor, Study Chair — Danish Research Centre for Cancer Diagnosis in Primary Care, Aarhus University, Denmark
Locations (1):
- Department of Molecular Medicine, Aarhus N, Aarhus, Denmark

REFERENCES:
- [Background] Fredsoe J, Kirkegaard P, Edwards A, Vedsted P, Sorensen KD, Bro F. A genetic risk assessment for prostate cancer influences patients' risk perception and use of repeat PSA testing: a cross-sectional study in Danish general practice. BJGP Open. 2020 Jun 23;4(2):bjgpopen20X101039. doi: 10.3399/bjgpopen20X101039. Print 2020. PMID 32457098
- [Background] Fredsoe J, Koetsenruyter J, Vedsted P, Kirkegaard P, Vaeth M, Edwards A, Orntoft TF, Sorensen KD, Bro F. The effect of assessing genetic risk of prostate cancer on the use of PSA tests in primary care: A cluster randomized controlled trial. PLoS Med. 2020 Feb 7;17(2):e1003033. doi: 10.1371/journal.pmed.1003033. eCollection 2020 Feb. PMID 32032355
- [Background] Kirkegaard P, Edwards A, Nielsen TLO, Orntoft TF, Sorensen KD, Borre M, Bro F. Perceptions about screening for prostate cancer using genetic lifetime risk assessment: a qualitative study. BMC Fam Pract. 2018 Feb 17;19(1):32. doi: 10.1186/s12875-018-0717-6. PMID 29454309
- [Derived] Kirkegaard P, Vedsted P, Edwards A, Fenger-Gron M, Bro F. A cluster-randomised, parallel group, controlled intervention study of genetic prostate cancer risk assessment and use of PSA tests in general practice--the ProCaRis study: study protocol. BMJ Open. 2013 Mar 1;3(3):e002452. doi: 10.1136/bmjopen-2012-002452. PMID 23457331